CLINICAL TRIAL: NCT00417092
Title: Biventricular Pacing After Coronary Artery Bypass Grafting (BIVAC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UL 04-156
Record Dates: First submitted 2006-12-28; First posted 2006-12-29 (Estimated); Last update posted 2007-09-24 (Estimated); Status verified 2007-09

CONDITIONS: Cardiac Pacing,Artificial; Coronary Artery Bypass; Ventricular Function, Left
Keywords: coronary artery bypass grafting; reduced left ventricular function; postoperative pacing; cardiac resynchronization

INTERVENTIONS:
Procedure: Postoperative Pacing

SUMMARY:
The purpose of this study is to determine which pacing mode after coronary artery bypass grafting in patients with reduced left ventricular function is hemodynamically favorable.

DETAILED DESCRIPTION:
Patients with severely reduced left ventricular function undergoing coronary artery bypass grafting (CABG) are at an increased perioperative risk and often need prolonged postoperative treatment on intensive care units. A significant portion of these patients require postoperative pacing. Right ventricular pacing has been shown to be hemodynamically deleterious whereas biventricular pacing improves cardiac output in patients with severely reduced left ventricular function and bundle branch block. The purpose of this study is to compare DDD-right ventricular, DDD-biventricular and AAI pacing in CABG patients with an ejection fraction less than 40% in a prospective randomized setting.

ELIGIBILITY:
Inclusion Criteria:

* Elective or urgent coronary artery bypass grafting
* Preoperative ejection fraction less than 40%

Exclusion Criteria:

* Existing permanent pacemaker or ICD
* Concomitant valve surgery
* Preoperative cardiovascular instability requiring intubation or IABP use
* Chronic renal failure requiring dialysis
* Failure to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-12; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Duration of Intensive Care Treatment

SECONDARY OUTCOMES:
30 day mortality
Major adverse events
Duration of Hospital Stay
Hemodynamic parameters
Inotrope use
Atrial fibrillation
Ventricular tachycardia / ventricular fibrillation
Renal function
Stability of pacing wires

CONTACTS AND LOCATIONS:
Overall Officials: Uwe KH Wiegand, MD, Study Director — University Hospital Schlesig Holstein, Campus Luebeck, Medicine II, Luebeck, Germany
Locations (1):
- University Hospital Schleswig Holstein, Campus Luebeck, Cardiac Surgery, Lübeck, Schleswig-Holstein, Germany